CLINICAL TRIAL: NCT03953404
Title: Bedside Measurements of a Novel Biomarker SPLA2-IIA as a Marker of an Inflammatory Response and Predictor of Sepsis in Patients Meeting SIRS or qSOFA Criteria: a Pilot Study
Brief Title: POC SPLA2-IIA as a Biomarker for Sepsis and Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Luke's Hospital, Pennsylvania (Other)
Responsible Party: Principal Investigator, rebecca jeanmonod, Professor of Emergency Medicine, St. Luke's Hospital, Pennsylvania
Other Study IDs: SLIR 2019-23
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- septic shock
  Interventions: Diagnostic Test: SPLA2-IIA
- severe sepsis
  Interventions: Diagnostic Test: SPLA2-IIA
- sepsis
  Interventions: Diagnostic Test: SPLA2-IIA
- sirs positive, not septic
  Interventions: Diagnostic Test: SPLA2-IIA

INTERVENTIONS:
Diagnostic Test: SPLA2-IIA — bedside blood test

SUMMARY:
Septic shock is a major cause of morbidity and mortality. SIRS (systemic inflammatory response syndrome) can progress over hours to days to severe sepsis and septic shock. Currently, lactate levels are used to guide resuscitative efforts and have been shown to be a predictor of mortality independent of vital sign abnormalities (1). However, their use seems to be limited to trending in a given patient, and not for prognostic value of a single level (2). This is because there is significant overlap in lactate levels of individuals who progress to death and multisystem organ failure as compared to those who do not (2). Blood cultures are also extensively used to detect blood stream infection (BSI), but these are time consuming and are not immediately useful to clinicians caring for sick patients.

A biomarker that adequately distinguishes between patients at high risk for progression to severe sepsis/shock/death and those who will not would be helpful in the appropriate initiation of aggressive treatment and appropriate disposition of patients in clinical care. Previously, the investigators demonstrated that sPLA2-IIA detected by ELISA assay had a sensitivity of 87% and a specificity of 91% in detecting sepsis (3). Zeus Pharmaceuticals has developed a bedside point-of-care test measuring sPLA2-IIA in real time. The investigators propose to study this assay in terms of its discriminatory value in distinguishing between SIRS from non-infectious causes, sepsis, severe sepsis, and septic shock in a cohort of patients presenting to the emergency department at Anderson and Bethlehem campuses. The investigators propose to better define the threshold level for this marker assay as well as seek to establish its utility in a clinical population.

The investigators will take samples of blood from emergency department patients presenting who meet SIRS criteria or have a positive q-SOFA screen. The investigators will take subsequent samples of blood when lactate levels are redrawn as per St. Luke's sepsis protocol. After informed consent is obtained, blood specimens will be run in analyzer provided by Zeus for sPLA2-IIA. The investigators will record presence and quantity of sPLA2-IIA, as well as other markers of sepsis such as lactate, vital signs, blood cultures, and patient oriented outcomes (ie ICU days, organ dysfunction, and survival to discharge). Printouts from analyzer will be stored in locked cabinet, and remaining blood will be discarded. The data will then be compiled by the investigators at St. Luke's University Hospital. The results will be correlated with the patients' clinical progression to determine the biomarker's utility and cut-off values for predicting progression of SIRS.

As clear threshold levels for this marker have yet to be defined, the investigators would like to enroll patients meeting criteria until the investigators have enrolled 50 patients with septic shock. It is anticipated that, proportionally, this will lead to enrollment of 75-100 patients with severe sepsis, 100-150 patients with sepsis, and 100-150 patients meeting SIRS criteria who are not septic. This will help delineate if there is any value in this assay for distinguishing among the severity of sepsis pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* presenting to emergency department with positive sepsis screen including 2 SIRS criteria or positive q-sofa score regardless of reasons for positive screen

Exclusion Criteria:

* inability to consent or to have surrogate consent, identification after resuscitation or after blood has already been drawn, age less than 18, pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: emergency department patients with positive sepsis screens
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
level greater than 25ng | baseline
  threshold level of spla2-IIA
level greater than 25ng | 2 hours
  threshold level of spla2-IIA
level greater than 25ng | 24 hour lab draw
  threshold level of spla2-IIA

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke'S University Health Network, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No